CLINICAL TRIAL: NCT04085055
Title: Randomized Trial Comparing Fine Needle Biopsy Needles and Different Techniques for Endoscopic-guided Fine Needle Biopsy of Solid Pancreatic Mass Lesions
Brief Title: Fine Needle Biopsy of Solid Pancreatic Mass Lesions
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: AdventHealth (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Single Group | Masking: Triple | Purpose: Diagnostic
Other Study IDs: 1469116
Record Dates: First submitted 2019-09-09; First posted 2019-09-11 (Actual); Last update posted 2020-08-05 (Actual); Status verified 2020-08

CONDITIONS: Pancreatic Neoplasms
Keywords: pancreatic mass, pancreatic solid mass, pancreatic lesion
MeSH Terms: conditions — Pancreatic Neoplasms | interventions — Biopsy, Fine-Needle

STUDY DESIGN:
Intervention Model Description: This is a randomized trial comparing four types of FNB needles and three sampling techniques. Patients will be randomized to one of the four different FNB needles. All patients will then undergo FNB using the specified needle and all three sampling techniques (one pass per technique using the assigned needle).
Who Masked: Participant, Care Provider, Outcomes Assessor
Masking Description: The patients, pathologists assessing the biopsy specimens and the research staff responsible for follow-up will be blinded to the FNB needle type utilized. Data will also be blinded for statistical analysis.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: Yes

ARMS (4):
- 22 Gauge FNB Needle - ProCore (Active Comparator): The 22 Gauge FNB Needle - ProCore will be used to biopsy solid pancreatic mass lesions.
  Interventions: Diagnostic Test: Solid pancreatic mass lesion biopsy
- 22 Gauge FNB Needle - Acquire (Active Comparator): The 22 Gauge FNB Needle - Acquire will be used to biopsy solid pancreatic mass lesions.
  Interventions: Diagnostic Test: Solid pancreatic mass lesion biopsy
- 22 Gauge FNB Needle - SharkCore (Active Comparator): The 22 Gauge FNB Needle - SharkCore will be used to biopsy solid pancreatic mass lesions.
  Interventions: Diagnostic Test: Solid pancreatic mass lesion biopsy
- 22 Gauge FNB needle - EZ Shot 3 Plus (Active Comparator): The 22 Gauge FNB Needle - EZ Shot 3 Plus will be used to biopsy solid pancreatic mass lesions.
  Interventions: Diagnostic Test: Solid pancreatic mass lesion biopsy

INTERVENTIONS:
Diagnostic Test: Solid pancreatic mass lesion biopsy — The needle will be used to puncture the lesion and remove a piece of tissue from the mass for histological diagnosis.
  Other Names: biopsy, fine needle biopsy, fine needle aspiration

SUMMARY:
This is a randomized trial to evaluate and directly compare the tissue quality, diagnostic sucess and safety profile of four different Fine Needle Biopsy needles.

DETAILED DESCRIPTION:
Endoscopic ultrasound-guided fine needle aspiration (EUS-FNA) is currently the standard method for sampling solid pancreatic masses, with reported sensitivity for malignant cytology of 85-95%, specificity of 95-98% and diagnostic accuracy of 78-95%. Diagnostic failure of EUS-FNA can be due to inadequate targeting, inexperience of the endoscopist/pathologist, or necrotic or fibrotic tumors in which viable cells are difficult to obtain. The cellularity and architectural representation of the sample can also be determined by the needle used and its specific features. Recently, new needles known as "fine needle biopsy (FNB)" needles have become available that are specially designed to promote the collection of core tissue by unique designs of their needle tips. The advantages of FNB over FNA needles are that (a) the quality of tissue procured is superior: FNA needles yield cytology whereas FNB needles yield histology (b) molecular marker analysis can be performed more reliably on histology samples than cytology aspirates and (c) as histological tissue is greater in quantity than cytological aspirates, a quicker diagnosis with fewer passes can be established by histology than cytology.

Four different types of FNB needles are currently available - reverse-bevel tip (EchoTip ProCore HD Ultrasound Biopsy Needle, Cook Medical, Bloomington, IN), Menghini-tip (EZ shot, Olympus America, Center Valley, PA), Franseen tip (Acquire, Boston Scientific Corporation, Natick, MA) and fork-tip (SharkCore, Medtronic Corporation/Covidien, Newton, MA) needles, each with unique tip designs to facilitate procurement of histological core tissue. Although we have previously compared in randomized trials the diagnostic yield of Franseen and fork-tip FNB needles and have shown the two needles to be equivalent, there are currently no randomized trials directly comparing all four FNB needle types. EUS-guided tissue acquisition can also be performed using different techniques, including the use of suction, no use of suction and the stylet retraction technique. There are currently no studies comparing these different tissue acquisition techniques using the different FNB needles and no study has demonstrated the best technique for FNB.

ELIGIBILITY:
Inclusion Criteria:

1. All patients referred for EUS-guided tissue acquisition of suspected or confirmed solid pancreatic mass lesions visualized on any radiological imaging
2. Able and willing to provide written or verbal consent
3. ≥ 18 years old
4. Able to undergo conscious sedation for EUS procedure

Exclusion Criteria:

1. <18 years old
2. Unable to obtain informed consent from the patient
3. Medically unfit for sedation
4. Pregnant patients
5. No pancreatic mass lesions visualized on EUS
6. Irreversible coagulopathy as determined by platelet count < 50,000/microL or International Normalized Ratio (INR) > 1.5
7. Unable to stop anti-platelet agents prior to the procedure

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 130 (Estimated)
Dates: Start 2019-09-09 (Actual); Primary Completion 2020-06-25 (Actual); Study Completion 2020-12 (Estimated)

PRIMARY OUTCOMES:
Degree of cellularity in biopsy sample | 3 days
  Compare the degree of cellularity of the obtained tissue in the biopsy sample between the four FNB needles in patients undergoing EUS-guided sampling of pancreatic masses using the three different sampling techniques. Cellularity is defined as the proportion of core tissue to total specimen area.

SECONDARY OUTCOMES:
Diagnostic adequacy of the biopsy sample | 1 day
  Documentation of the presence of adequate tissue material (pancreatic parenchyma and tumor if applicable) in the biopsy sample.
Specimen bloodiness in biopsy sample | 1 day
  Measured as the area of bloodiness in the biopsy sample, with calculation as a percentage in the microscopic field.
Presence of crush artefact in biopsy sample | 1 day
  Documenting the presence or absence of crush artefact in the biopsy sample. If present, it is measured as the area of artefact in biopsy sample, with calculation as a percentage in relation to the total sample area.
Technical failure | 1 day
  Measured as the inability to successfully perform the fine needle biopsy using the assigned needle, due to any needle dysfunction.
Adverse events | 7 days, 30 days, and 6 months
  The subject will be asked to report and medical records will be reviewed for any adverse events related to the procedure or the underlying disease.
Diagnostic operating characteristics | 6 months
  Compare the diagnostic operating characteristics of the biopsy sample and detection of neoplasia (defined as sensitivity, specificity, negative predictive value, positive predictive value and accuracy) between the four FNB needles in patients undergoing EUS-guided sampling of pancreatic masses using the three different sampling techniques

CONTACTS AND LOCATIONS:
Overall Officials: Shyam Varadarajulu, MD, Principal Investigator — AdventHealth
Locations (1):
- AdventHealth Orlando, Orlando, Florida, United States

REFERENCES:
- [Background] Ngamruengphong S, Li F, Zhou Y, Chak A, Cooper GS, Das A. EUS and survival in patients with pancreatic cancer: a population-based study. Gastrointest Endosc. 2010 Jul;72(1):78-83, 83.e1-2. doi: 10.1016/j.gie.2010.01.072. PMID 20620274
- [Background] Othman MO, Wallace MB. The role of endoscopic ultrasonography in the diagnosis and management of pancreatic cancer. Gastroenterol Clin North Am. 2012 Mar;41(1):179-88. doi: 10.1016/j.gtc.2011.12.014. Epub 2012 Jan 16. PMID 22341257
- [Background] Hewitt MJ, McPhail MJ, Possamai L, Dhar A, Vlavianos P, Monahan KJ. EUS-guided FNA for diagnosis of solid pancreatic neoplasms: a meta-analysis. Gastrointest Endosc. 2012 Feb;75(2):319-31. doi: 10.1016/j.gie.2011.08.049. PMID 22248600
- [Background] Varadarajulu S, Fraig M, Schmulewitz N, Roberts S, Wildi S, Hawes RH, Hoffman BJ, Wallace MB. Comparison of EUS-guided 19-gauge Trucut needle biopsy with EUS-guided fine-needle aspiration. Endoscopy. 2004 May;36(5):397-401. doi: 10.1055/s-2004-814316. PMID 15100946
- [Background] Bang JY, Hawes R, Varadarajulu S. A meta-analysis comparing ProCore and standard fine-needle aspiration needles for endoscopic ultrasound-guided tissue acquisition. Endoscopy. 2016 Apr;48(4):339-49. doi: 10.1055/s-0034-1393354. Epub 2015 Nov 12. PMID 26561917
- [Background] Bang JY, Hebert-Magee S, Navaneethan U, Hasan MK, Hawes R, Varadarajulu S. EUS-guided fine needle biopsy of pancreatic masses can yield true histology. Gut. 2018 Dec;67(12):2081-2084. doi: 10.1136/gutjnl-2017-315154. Epub 2017 Oct 7. No abstract available. PMID 28988195
- [Background] Bang JY, Hebert-Magee S, Navaneethan U, Hasan MK, Hawes R, Varadarajulu S. Randomized trial comparing the Franseen and Fork-tip needles for EUS-guided fine-needle biopsy sampling of solid pancreatic mass lesions. Gastrointest Endosc. 2018 Jun;87(6):1432-1438. doi: 10.1016/j.gie.2017.11.036. Epub 2018 Jan 3. PMID 29305893
- [Background] Lee KY, Cho HD, Hwangbo Y, Yang JK, Han SJ, Choi HJ, Lee YN, Cha SW, Moon JH, Cho YD, Park SH, Lee TH. Efficacy of 3 fine-needle biopsy techniques for suspected pancreatic malignancies in the absence of an on-site cytopathologist. Gastrointest Endosc. 2019 Apr;89(4):825-831.e1. doi: 10.1016/j.gie.2018.10.042. Epub 2018 Nov 4. PMID 30403966
- [Background] Saxena P, El Zein M, Stevens T, Abdelgelil A, Besharati S, Messallam A, Kumbhari V, Azola A, Brainard J, Shin EJ, Lennon AM, Canto MI, Singh VK, Khashab MA. Stylet slow-pull versus standard suction for endoscopic ultrasound-guided fine-needle aspiration of solid pancreatic lesions: a multicenter randomized trial. Endoscopy. 2018 May;50(5):497-504. doi: 10.1055/s-0043-122381. Epub 2017 Dec 22. PMID 29272906
- [Background] Nakai Y, Isayama H, Chang KJ, Yamamoto N, Hamada T, Uchino R, Mizuno S, Miyabayashi K, Yamamoto K, Kawakubo K, Kogure H, Sasaki T, Hirano K, Tanaka M, Tada M, Fukayama M, Koike K. Slow pull versus suction in endoscopic ultrasound-guided fine-needle aspiration of pancreatic solid masses. Dig Dis Sci. 2014 Jul;59(7):1578-85. doi: 10.1007/s10620-013-3019-9. Epub 2014 Jan 16. PMID 24429514
- [Background] Chow, S.C.; Shao, J.; Wang, H. 2008. Sample Size Calculations in Clinical Research, 2nd Edition. Chapman & Hall/CRC. Boca Raton, FL. Pages 99-100.
- [Derived] Young Bang J, Krall K, Jhala N, Singh C, Tejani M, Arnoletti JP, Navaneethan U, Hawes R, Varadarajulu S. Comparing Needles and Methods of Endoscopic Ultrasound-Guided Fine-Needle Biopsy to Optimize Specimen Quality and Diagnostic Accuracy for Patients With Pancreatic Masses in a Randomized Trial. Clin Gastroenterol Hepatol. 2021 Apr;19(4):825-835.e7. doi: 10.1016/j.cgh.2020.06.042. Epub 2020 Jul 8. PMID 32652307